CLINICAL TRIAL: NCT06639074
Title: MC1963 Folate Receptor Alpha Dendritic Cells (FRαDCs) or Placebo for Patients With Advanced Stage Ovarian Cancer: A Phase II Double-Blind Randomized Clinical Trial (FAROUT)
Brief Title: Folate Receptor Alpha Dendritic Cells (FRαDCs) or Placebo for the Treatment of Patients With Stage III or IV Ovarian, Fallopian Tube, or Primary Peritoneal Cancer, FAROUT Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MC1963; NCI-2024-08466 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-000088 (Other: Mayo Clinic Institutional Review Board); MC1963 (Other: Mayo Clinic)
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Advanced Fallopian Tube Carcinoma; Advanced Fallopian Tube High Grade Serous Adenocarcinoma; Advanced Ovarian Carcinoma; Advanced Ovarian Carcinosarcoma; Advanced Ovarian Clear Cell Adenocarcinoma; Advanced Ovarian Endometrioid Adenocarcinoma; Advanced Ovarian High Grade Serous Adenocarcinoma; Advanced Primary Peritoneal Carcinoma; Advanced Primary Peritoneal High Grade Serous Adenocarcinoma; Fallopian Tube Carcinosarcoma; Fallopian Tube Clear Cell Adenocarcinoma; Fallopian Tube Endometrioid Adenocarcinoma; FIGO Stage III Ovarian Cancer 2014; FIGO Stage IV Ovarian Cancer 2014; Ovarian Mixed Cell Adenocarcinoma; Primary Peritoneal Carcinosarcoma; Primary Peritoneal Clear Cell Adenocarcinoma; Primary Peritoneal Endometrioid Adenocarcinoma
MeSH Terms: interventions — Biopsy; Specimen Handling; Diphtheria Toxoid; adacel; Diphtheria-Tetanus-acellular Pertussis Vaccines; Tetanus Toxoid; Leukapheresis; Magnetic Resonance Spectroscopy; Diphtheria-Tetanus Vaccine

STUDY DESIGN:
Intervention Model Description: Participants are allocated randomly to vaccine versus placebo in a 2:1 fashion.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patient, provider and principal investigator are blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (FRalphaDCs) (Experimental): Patients may receive Td or Tdap IM prior to undergoing leukapheresis. Patients receive FRalphaDCs ID on day 1 of each cycle. Cycles repeat every 21 days for cycles 1-5 and then repeat every 91 days for cycles 6-12 in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo biopsy prior to apheresis and optionally at end of treatment, and blood sample collection, CT and/or MRI throughout the study.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Diphtheria Toxoid/Tetanus Toxoid/Acellular Pertussis Vaccine Adsorbed; Procedure: Leukapheresis; Procedure: Magnetic Resonance Imaging; Biological: Multi-epitope Folate Receptor Alpha-loaded Dendritic Cell Vaccine; Biological: Tetanus and Diphtheria Toxoids Adsorbed
- Arm II (placebo) (Placebo Comparator): Patients may receive Td or Tdap IM prior to undergoing leukapheresis. Patients receive placebo ID on day 1 of each cycle. Cycles repeat every 21 days for cycles 1-5 and then repeat every 91 days for cycles 6-12 in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo biopsy prior to apheresis and optionally at end of treatment, and blood sample collection, CT and/or MRI throughout the study.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Diphtheria Toxoid/Tetanus Toxoid/Acellular Pertussis Vaccine Adsorbed; Procedure: Leukapheresis; Procedure: Magnetic Resonance Imaging; Drug: Placebo Administration; Biological: Tetanus and Diphtheria Toxoids Adsorbed

INTERVENTIONS:
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Biological: Diphtheria Toxoid/Tetanus Toxoid/Acellular Pertussis Vaccine Adsorbed — Given IM
  Other Names: Adacel; Daptacel; Diphtheria and Tetanus Toxoids and Acellular Pertussis Vaccine Adsorbed; Diphtheria Toxoid Tetanus Toxoid Acellular Pertussis Vaccine Adsorbed; Diphtheria Toxoid/Tetanus Toxoid/Acellular Pertussis Vaccine; DTaP; Infanrix; Tripedia
Procedure: Leukapheresis — Undergo leukapheresis
  Other Names: Leukocyte Adsorptive Apheresis; Leukocytopheresis; Therapeutic Leukopheresis; White Blood Cell Reduction Apheresis
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Multi-epitope Folate Receptor Alpha-loaded Dendritic Cell Vaccine — Given ID
  Other Names: FRaDC Vaccine; FRalphaDC Vaccine
  Arms: Arm I (FRalphaDCs)
Drug: Placebo Administration — Given ID
  Arms: Arm II (placebo)
Biological: Tetanus and Diphtheria Toxoids Adsorbed — Given IM
  Other Names: DECAVAC; Td; Tetanus and Diphtheria Toxoids Adsorbed for Adult Use

SUMMARY:
This phase II trial compares the effect of folate receptor alpha dendritic cells (FRαDCs) to placebo in treating patients with stage III or IV ovarian, fallopian tube or primary peritoneal cancer. FRαDCs, a dendritic cell vaccine, is made from a person's white blood cells. The white blood cells are treated in the laboratory to make dendritic cells (a type of immune cell) mixed with folate receptor alpha (FRalpha), a protein found in high levels on ovarian tumor cells. FRαDCs work by boosting the immune system to recognize and destroy the tumor cells by targeting the FRalpha protein on the tumor cell. Placebo is an inactive substance that looks the same as, and is given the same way as, the active drug or treatment being tested. The effects of the active drug are compared to the effects of the placebo. Giving FRαDCs may work better in preventing or delaying recurrence compared to placebo in patients with stage III or IV ovarian, fallopian tube, or primary peritoneal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Compare recurrence-free survival (RFS) in advanced ovarian carcinoma (OC) patients vaccinated with multi-epitope folate receptor alpha-loaded dendritic cell vaccine (FRαDCs) (active vaccine) versus placebo.

SECONDARY OBJECTIVES:

I. Compare overall survival (OS) in advanced OC patients vaccinated with FRαDCs versus placebo.

II. Compare the adverse event (AE) profile of FRαDCs with that of placebo.

CORRELATIVE RESEARCH OBJECTIVES:

I. Assess association of pre-existing immune microenvironment with RFS. II. Characterize the T cell and antibody responses to FRα and assess the association between the emergence of immunity and RFS.

III. Assess for epitope spreading and evaluate the association between epitope spreading and RFS.

IV. Compare archival tissue from surgery with post-recurrence biopsy tissue in those patients who develop recurrence to assess for common immune evasion mechanisms.

V. Evaluate differences in ribonucleic acid (RNA) expression of FRαDCs and its association with RFS.

OUTLINE: Patients are randomized to 1 of 2 arms. Randomization is 2:1, vaccine to placebo.

ARM I: Patients may receive tetanus and diphtheria vaccine (Td) or tetanus-diphtheria-accellular pertussis vaccine (Tdap) intramuscularly (IM) prior to undergoing leukapheresis. Patients receive FRalphaDCs intradermally (ID) on day 1 of each cycle. Cycles repeat every 21 days for cycles 1-5 and then repeat every 91 days for cycles 6-12 in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo biopsy prior to apheresis and optionally at end of treatment, and blood sample collection, computed tomography (CT) and/or magnetic resonance imaging (MRI) throughout the study.f

ARM II: Patients may receive Td or Tdap IM prior to undergoing leukapheresis. Patients receive placebo ID on day 1 of each cycle. Cycles repeat every 21 days for cycles 1-5 and then repeat every 91 days for cycles 6-12 in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo biopsy prior to apheresis and optionally at end of treatment, and blood sample collection, CT and/or MRI throughout the study.

After completion of study treatment, patients are followed up every 3 months for up to month 36 then every 3 months until progression followed by every 6 months for up to year 8.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histological confirmation of Federation of Gynecology and Obstetrics (FIGO) stage III or stage IV epithelial ovarian, fallopian tube, or primary peritoneal cancer. NOTE: Histologic confirmation of the primary tumor is required. Eligible histotypes include high grade serous; endometrioid; and clear cell carcinoma, as these histotypes have high expression of FRα (Kalli, Oberg, Keeney, & et al., 2008). Mixed carcinomas, including carcinosarcomas, with ≥ 50% of the tumor comprised of high grade serous; and/or endometrioid; and/or clear cell carcinoma are eligible
* Completion of cytoreductive surgery and one (and only one) course of platinum-based chemotherapy (5-9 cycles) ≥ 4 but ≤ 12 weeks prior to registration

  * NOTE: Cytoreductive surgery may have been prior to or after one or more cycles of chemotherapy and must include hysterectomy and bilateral salpingo-oophorectomy (if the uterus and/or ovaries were not previously removed)
  * NOTE: Patients may have had more than one chemotherapy regimen (examples: paclitaxel/carboplatin switched to docetaxel/carboplatin due to allergy; or weekly treatment switched to every 3-weekly treatment due to intolerance), but may not have received a separate course of treatment for recurrent OC
  * NOTE: Patients may receive both neoadjuvant and adjuvant chemotherapy provided both regimens are platinum-based and total nine (9) or fewer chemotherapy cycles
* Germline and somatic genetic testing have been completed

  * NOTE: No pathogenic mutations of BRCA1/BRCA2 are allowed
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, or 2
* Expected survival ≥ 6 months
* Hemoglobin ≥ 8.5 g/dL (≤ 15 days prior to registration)
* Absolute neutrophil count (ANC) ≥ 1000/mm^3 (≤ 15 days prior to registration)
* Platelet count ≥ 75,000/mm^3 (≤ 15 days prior to registration)
* Lymphocytes ≥ 0.3 x 10^9/L (≤ 15 days prior to registration)
* Monocytes ≥ 0.25 x 10^9/L (≤ 15 days prior to registration)
* Total bilirubin ≤ upper limit of normal (ULN), unless patient has a documented history of Gilbert's disease, then direct bilirubin ≤ ULN (≤ 15 days prior to registration)
* Aspartate transaminase (AST) ≤ 3 x ULN (≤ 15 days prior to registration)
* Creatinine clearance ≥ 30 mL/min per Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) creatinine equation (≤ 15 days prior to registration)
* Provide written informed consent
* Willing to provide mandatory blood specimens for correlative research
* Willing to provide archival tissue specimen for correlative research
* Willing to return a participating institution for follow-up (during the active monitoring phase of the study)
* Willing to undergo a tetanus vaccination (if not performed ≤ 365 days prior to registration)
* Willing to have a central access line placed, if needed (as determined during venous access assessment)

Exclusion Criteria:

* Any of the following because this study involves an investigational agent, the genotoxic, mutagenic, and teratogenic effects of which on the developing fetus and newborn are unknown

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential or able to father a child who are unwilling to employ adequate contraception
* Evidence of disease at the time of registration, including clinical concern for disease recurrence based on each of the following:

  * Evidence of disease by history and physical exam
  * CA125 outside institutional normal limits
  * CT (and or MRI) of the chest/abdomen/pelvis demonstrating radiological evidence of disease performed after completion of chemotherapy ≤ 28 days be-fore entering study
* Germline or somatic BRCA1 or BRCA2 mutation, as determined by Clinical Laboratory Improvement Act (CLIA)-approved tests
* Prior radiation therapy for this cancer
* Treatment with chemotherapy, angiogenesis inhibitor therapy, poly (ADP-ribose) polymerase (PARP) inhibitor therapy, radiation therapy, or other immunotherapy ≤ 4 weeks prior to registration
* Receiving any other standard therapy (angiogenesis inhibitor, PARP inhibitor) or investigational agent, which would be considered as a treatment for the primary neoplasm. These agents have been shown to be active in later line therapy and can be used at that time for patients who relapse after treatment on this trial
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Immunocompromised patients and patients known to be HIV positive and currently receiving antiretroviral therapy

  * NOTE: Patients known to be HIV positive, but without clinical evidence of an immunocompromised state, are eligible for this trial
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study requirements
  * EXCEPTIONS: HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial. For patients with evidence of hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated. Patients with a history of hepatitis C virus (HCV) must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Other active malignancy ≤ 3 years prior to registration

  * EXCEPTIONS: Patients with non-melanotic skin cancer, papillary thyroid cancer not requiring therapy or carcinoma-in-situ are eligible for this trial. Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial. (Contact site principal investigator [PI] if questions.)
* History of myocardial infarction ≤ 6 months prior to registration, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias

  * NOTE: Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* Treatment with systemic immunosuppressive medication (including, but not limited to, prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [TNF]-alpha agents) ≤ 2 weeks prior to registration, or anticipation of need for systemic immunosuppressive medication during the course of the study

  * NOTE: Patients who have received acute, low-dose systemic steroids (≤ 10 mg/day oral prednisone or equivalent) prior to registration or a one-time pulse dose of systemic immunosuppressant medication (e.g., ≤ 48 hours of corticosteroids for a contrast allergy) are eligible for the study
  * NOTE: The use of inhaled corticosteroids for chronic obstructive pulmonary disease or asthma, mineralocorticoids (e.g., fludrocortisone), or low-dose corticosteroids for patients with orthostatic hypotension or adrenocortical insufficiency is allowed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-11-08 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival | Up to 8 years
  Recurrence-free survival (RFS) will be compared inadvanced OC patients vaccinated with FRαDCs (active vaccine) versus placebo. RFS is defined as the time from study entry to either disease recurrence or death from any cause.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 8 years
  Overall survival (OS) will be compared in advanced OC patients vaccinated with FRαDCs versus placebo. OS is defined as the time from study entry to death from any cause.
Incidence of adverse events (AEs) | Up to 30 days after last dose of study treatment
  The maximum grade for each type of AE will be summarized using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The frequency and percentage of grade 3 and greater AEs will be compared between the 2 arms.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew S. Block, MD, PhD, Principal Investigator — Mayo Clinic in Rochester
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials